CLINICAL TRIAL: NCT05217420
Title: Moving Well Intervention for Patients Preparing to Undergo Total Knee Arthroplasty (TKA)
Brief Title: Moving Well for Total Knee Arthroplasty (TKA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Rheumatology Research Foundation (Other); Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-08020638
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: arthroplasty; replacement; peer coach
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only research team members who will collect objective in-person data will be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moving Well (Experimental): Participants will receive weekly calls for 12 weeks (7 weeks before total knee arthroplasty surgery and 5 weeks after surgery) from a peer coach, an exercise program, and mental preparation (through positive thinking) for surgery. Participants will also receive the standard of care for patients undergoing total knee arthroplasty.
  Interventions: Behavioral: Moving Well
- Staying Well (Active Comparator): Participants will receive weekly calls for 12 weeks (7 weeks before total knee arthroplasty surgery and 5 weeks after surgery) from a research assistant. The calls will be similar in length to those in the experimental arm and will cover various health topics not related to total knee arthroplasty. Participants will also receive the standard of care for patients undergoing total knee arthroplasty.
  Interventions: Behavioral: Staying Well

INTERVENTIONS:
Behavioral: Moving Well — Experimental arm
  Arms: Moving Well
Behavioral: Staying Well — Active comparator arm
  Arms: Staying Well

SUMMARY:
The purpose of this study is to assess the efficacy of a behavioral intervention, Moving Well, in improving levels of anxiety and depression for patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Moving Well is a behavioral intervention, guided by peer coaches, that aims to improve mental and physical preparation for patients planning to undergo total knee arthroplasty (TKA) and improve postoperative recovery and outcomes. Peer coaches are patients who themselves have had TKA due to advanced osteoarthritis (OA) of the knee and have been trained and certified to become peer coaches.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have their primary TKR (one knee or both knees) scheduled in 8 weeks or more
* Be willing to participate in the Moving Well (intervention) arm or Staying Well (attention control) arm
* Are willing to work with a coach
* ≥ 50 years of age
* Speak English
* Have access to the internet, computer, and a working phone
* We will prioritize the recruitment of subjects with low socioeconomic status defined as being a beneficiary of Medicaid or no insurance and an underrepresented racial/ethnic group (Hispanic/Black).

Exclusion Criteria:

* Non-English speakers
* The intervention will first be delivered in English to ensure feasibility with the content before adapting the material for patients who speak other languages.
* TKR was a result of a septic joint or revision (implant malfunction)
* Unable to exercise (e.g., bed bound or wheelchair bound)
* Have had contralateral TKR or other joint replacement surgery (hip, shoulder) within the past 5 years
* If they have RA or other connective tissue disease: Lupus, ankylosing spondylitis, psoriatic arthritis, scleroderma, infectious arthritis, polymyalgia rheumatica.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in level of anxiety from baseline using the Generalized Anxiety Disorder Assessment (GAD-7) | Baseline, 6 months post-surgery
  The GAD-7 is a 7 item self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. Scores range from 0 to 21, with higher scores indicating greater severity of anxiety.
Change in level of depression from baseline using the Patient Health Questionnaire-8 (PHQ-8) | Baseline, 6 months post-surgery
  The PHQ-8 is a 8 item scale that screens for depression. Scores range from 0 to 24 with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Change in level of social support from baseline using the Lubben Social Network Scale-18 (LSNS-18) | Baseline, 6 months post-surgery
  The LSNS-18 is a 18 item scale that measures perceived social support. Scores range from 0 to 90 with higher scores indicating greater social engagement.
Change in general health status from baseline using the 12-Item Short Form Survey (SF-12) | Baseline, 6 months post-surgery
  The SF-12 is a 12 item scale that assesses general health status. Scores range from 0 to 100 with higher scores indicating better physical and mental health functioning.
Change in level of pain catastrophizing from baseline using the Pain Catastrophizing Scale (PCS). | Baseline, 6 months post-surgery
  The PCS is a 13 item scale that assesses the level of catastrophic thinking related to an individual's pain. Scores range from 0 to 52 with higher scores indicating a higher level of pain-related anxiety.
Change in level of knee pain and function from baseline using the Knee Injury and Osteoarthritis Outcome Score (KOOS) pain sub-scale. | Baseline, 6 months post-surgery
  The KOOS pain sub-scale is a 9 item scale that assesses knee pain. Scores range from 0 to 100 with lower scores indicating greater severity of pain. The KOOS function sub-scale is a 17 item scale that assesses function. Scores range from 0 to 100 with lower scores indicating worse knee function.
Change in level of self-efficacy from baseline using the General Self-Efficacy Scale (GSF) | Baseline, 6 months post-surgery
  The GSF is a 10 item scale that assesses perceived self-efficacy. Scores range from 10 to 40 with higher scores indicating a higher level of self-efficacy.
Change in sleep disturbance from baseline using the Patient-Reported Outcomes Information System (PROMIS) Sleep Disturbance Scale. | Baseline, 6 months post-surgery
  The PROMIS Sleep Disturbance Scale is a 8 item scale that measure self-reported perceptions of sleep quality, depth, and restoration within the past seven days. Scores range from with higher scores indicating greater sleep disturbances.
Change in opioid use for knee pain from baseline using participant self-report | Baseline, 6 months post-surgery
  Self-reported use of opioids for knee pain
Duration of post-surgery inpatient rehabilitation using the number of days of inpatient rehabilitation | 6 months post-surgery
  Self-reported duration of inpatient rehabilitation
Change in knee range of motion from baseline using a goniometer | Baseline, 6 months post-surgery
  A goniometer measures the range of motion at a joint. Measurement ranges from 0 to 180 degrees with higher range indicating greater range of motion.
Change in Timed Up and Go test (TUG) from baseline | Baseline, 6 months post-surgery
  The Timed Up and Go test is used to assess mobility. Completing the test in more than 12 seconds indicates a greater risk of falling in older adults.
Change in 6-minute walk test (6MWT) from baseline | Baseline, 6 months post-surgery
  The 6MWT is used to assess aerobic capacity and endurance. The distance covered by walking for 6 minutes is measured and used to compare changes in performance capacity.
Change in 30-second chair to stand test from baseline | Baseline, 6 months post-surgery
  The 30-second chair to stand test assesses leg strength and endurance. Scoring is based on the number of stands with a lower than average number indicating a greater risk of falls.
Change in quadriceps strength from baseline using a handheld dynamometer (HHD) | Baseline, 6 months post-surgery
  A handheld dynamometer is a device that measures muscle strength. Scores range from 0-300 pounds (upper limit can vary based on the device) with higher scores indicating greater quadriceps muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Y Navarro Millan, MD, MSPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine Clinical & Translational Science Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jabri A, Dominguez Paez Y, Brown M, Lui G, Hui WK, Hernandez N, Parks ML, Gonzalez Della Valle A, Goodman SM, Banerjee S, Safford MM, Navarro-Millan I. A single-center, open-label, randomized, parallel-group trial to pilot the effectiveness of a peer coach behavioral intervention versus an active control in reducing anxiety and depression in patients scheduled for total knee replacement. BMC Musculoskelet Disord. 2023 May 5;24(1):353. doi: 10.1186/s12891-023-06460-4. PMID 37147587